CLINICAL TRIAL: NCT06088147
Title: Methotrexate With Microneedling Versus Triamcinilone Acetonide With Microneedling in Treatment of Recalcitrant Alopecia Areata
Brief Title: Methotrexate Versus Triamcinilone Acetonide in Treatment of Recalcitrant Alopecia Areata
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Athar Fathy Abodief, Doctor, Al-Azhar University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSc/AZ.AST/DVA021/6/215/1/2023
Record Dates: First submitted 2023-08-25; First posted 2023-10-18 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Alopecia Areata
Keywords: Alopecia areata; Methotrexate; Triamcinolone; microneedling
MeSH Terms: conditions — Alopecia Areata | interventions — Methotrexate; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1= Methotrexate (Active Comparator): After microneedling, we will apply methotrexate topically (25 mg/ml) on half of the scalp at a dose of 0.02ml/cm2 with a maximum of 0.1-0.2 ml (2,5-5 mg) and rub it gently. The patient will take a session every 2 weeks for 12 weeks, on the same patient on the other patch or half of the scalp according to the pattern.
  Interventions: Drug: Methotrexate
- Group2=Triamcinilone (Experimental): we will use Triamcinolone acetonide 40 mg/1ml after microneedking at dose 5mg/ml concentration;1/8/ 1:7 dilution session every 3 weeks for 12 weeks. then after 12 weeks of treatment we will follow up our patients after discontinuing therapy for other 12 weeks and evaluate.
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Methotrexate — A standard derma pen 12 pins with of 0,5 mm depth was used, dermapen as a tool of infusion of our treatments works in a few ways to target hair loss, firstly by breaking down the scar tissue that covers or compromises the hair follicles which are not growing, stimulating new hair growth and also by enhancing infusion of mesotherapy ingredients to increase hair follicle size and therefore hair volume ,here we will use it by stamping technique, the procedure was practically painless and therefore no local anesthesia was used, however For those who will not want to tolerate pain, topical anesthesia with 2% lignocaine, under occlusion will applied, the patients will be followed up for 6 months after full course of treatment. Then we will apply methotrexate topically (25 mg/ml) on half of the scalp at a dose of 0.02ml/cm2
  Arms: Group 1= Methotrexate
Drug: Triamcinolone Acetonide — A standard derma pen 12 pins with of 0,5 mm depth was used, will use it by stamping technique, the procedure was practically painless and therefore no local anesthesia was used, however For those who will not want to tolerate pain, topical anesthesia with 2% lignocaine, under occlusion will applied, the patients will be followed up for 6 months after full course of treatment. Then Triamcinolone acetonide 40 mg/1ml after microneedking at dose 5mg/ml concentration;1/8/ 1:7 dilution
  Arms: Group2=Triamcinilone

SUMMARY:
Alopecia areata is the second most common cause of hair loss following androgenic alopecia.

It is affecting 2% of global population with an increasing prevalence. Briefly, it is a chronic, immunomediated disease characterized by acute onset of non-scarring hair loss ranging from small circumscribed patchy areas on the scalp to complete scalp and body hair loss. Until recently our understanding of the pathophysiology of alopecia areata is scarce, despite being so common.

Methotrexate is an immunosuppressant drug that has been widely used for a range of inflammatory and immune-mediated skin disorders.

Methotrexate has been recently proven to inhibit Jak/STAT Pathway. Triamcinolone acetonide as another type of treatment of alopecia areata either intralesionally or topically remains the first line of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age groups: > 12 years old.
* Sex: both sexes.
* Co-operative Patients.
* Recalcitrant or resistant cases to treatment (meaning that all patients had received various modalities of treatment in the past with poor/partial response or relapse after discontinuing therapy.

Exclusion Criteria:

* Patients <12 years.
* Pregnant and lactating women.
* Patients with any underlying Systemic disorders.
* Patients with HBV or HCV.
* Patient with active infection of T.B.
* Patients with bone marrow suppression (leukopenia, thrombocytopenia)
* Patients who had received any other modalities of treatment in last 3-6 months.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — microneedling is a painful technique so patients <12 years will be excluded
Enrollment: 34 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of methotrexate with microneedling versus triamcinolone with microneedling in treatment of recalcitrant alopecia areata. | 6 months
  Mcdonald Hull and Norris regrowth scale by trichoscope (Time frame 6 months). Grade 1: Regrowth of vellus hair, Grade 2: Regrowth of sparse pigmented terminal hair (<50% increment in % SALT score according to NAAF guideline), Grade 3: regrowth of terminal hair with patches of alopecia (50-75% increase in % SALT score), Grade 4: regrowth of terminal hair on the whole alopecia patch (> 75% increase in% SALT score).

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided